CLINICAL TRIAL: NCT02754011
Title: Dose-escalation, Phase I Multicentric Trial, Evaluating the Combination of Ribociclib and Capecitabine in Locally Advanced or Metastatic Breast Cancer HER2 Negative in Patients Previously Treated With Anthracyclines and Taxanes
Brief Title: Phase I Evaluating the Combination of Ribociclib+Capecitabine in Locally Advanced/Metastatic Breast Cancer HER2 Negative
Acronym: GEP14-LEECAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0101/1504
Record Dates: First submitted 2016-02-19; First posted 2016-04-28 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: HER2 negative; Locally advanced or metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination of ribociclib + capecitabine (Experimental): RIBOCICLIB from 200 to 600mg once daily + CAPECITABINE from 750 to 1000 mg/m² BID, cycles are defined in 21-day periods, 2 weeks on treatment, 1 week off treatment
  Interventions: Drug: Combination of ribociclib + capecitabine

INTERVENTIONS:
Drug: Combination of ribociclib + capecitabine — RIBOCICLIB from 200 to 600mg once daily + CAPECITABINE from 750 to 1000 mg/m² BID, cycles are defined in 21-day periods, 2 weeks on treatment, 1 week off treatment
  Other Names: Combination of LEE011 and XELODA

SUMMARY:
The proposed study is a multicenter, open-label phase I trial, conducted in locally advanced or metastatic breast cancer HER2 negative patients and divided into 2 parts:

* STEP 1: a dose escalation part (n= up to 30) to evaluate the safety profile and pharmacokinetics and to define the MTD and RP2D to recommend in a phase II.
* STEP 2: an expansion cohort part to confirm the safety and tolerability of ribociclib and capecitabine association on a longer follow-up, and to obtain preliminary evidence of anti-tumor activity on two expanded cohorts of HR positive and HR negative patients. Up to 14 patients in each cohort, taking into account patients already included in step one at this DL, may be enrolled, for a total of 28 at the RP2D.

DETAILED DESCRIPTION:
Patients with HER2 negative locally advanced or metastatic breast cancer, eligible to a capecitabine treatment as required by its approved indication, i.e previously treated with anthracyclines and taxanes

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 or more
2. Histologically-confirmed advanced breast cancer (metastatic or locally advanced)
3. Progressive patients who are eligible to a treatment with capecitabine: after failure to taxanes (neoadjuvant, adjuvant or metastatic setting) and failure to prior anthracycline-based chemotherapy (unless contraindicated)
4. Tumor no overexpressing HER2 (HER2 1+ in IHC, or IHC 2+ and FISH/ CISH negative) in samples from the primary and/or secondary tumor
5. A representative tumor specimen must be available for future research programs. An archival tumor sample may be submitted; however, if one is not available, a newly obtained tumor biopsy specimen must be submitted instead
6. Measurable or evaluable disease according to RECIST v1.1 criteria
7. Patients must be able to swallow tablets and capsules
8. Patients must have an estimated survival of at least 3 months
9. WHO performance status (ECOG) from 0 to 1
10. Adequate hematological and coagulation function: Hb ≥ 9.0 g/dL, ANC ≥ 1500/mm³ platelets ≥ 100 000/mm³, INR ≤ 1.5
11. Adequate hepatic function: total bilirubin ≤ ULN, or total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN in patients with well documented Gilbert's Syndrome, ALAT and ASAT ≤ 2.5 x ULN (regardless of the presence or absence of liver metastasis)
12. Adequate renal function: serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min
13. Adequate ionic balance: potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
14. Women of child-bearing potential must agree to use an effective contraceptive method while on treatment and for 8 weeks after study drugs discontinuation. Highly effective contraception methods are detailed in section 6.1.1.
15. Patient must be affiliated to a Social Security system
16. Patient information and written informed consent form signed

Exclusion Criteria:

1. Patient has been pre-treated by CDK inhibitor or capecitabine
2. Patient has a DPD deficiency
3. Patient has a known hypersensitivity to to 5-FU or to any of the excipients of ribociclib or capecitabine
4. Patients with central nervous system (CNS) involvement unless they meet ALL of the following criteria:

   * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
   * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases
5. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
6. Patient has a known history of HIV infection (testing not mandatory)
7. Clinically significant, uncontrolled heart disease and/or recent events including any of the following:

   * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to screening
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
   * Patient has a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
   * History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening
   * Congenital long QT syndrome or family history of long QT syndrome
   * Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening
   * Bradycardia (heart rate <50 at rest), by ECG or pulse, at screening
8. On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF >450 msec (using Fridericia's correction). All as determined by screening ECG (mean of triplicate ECGs)
9. Patient is currently receiving any of the following medications (see Table 9 for details) and cannot be discontinued 7 days prior to starting study drugs:

   * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruits hybrids, pummelos, star-fruit, and Seville oranges
   * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
   * That have a known risk to prolong the QT interval or induce Torsades de Pointes
   * Herbal preparations/medications, dietary supplements
10. Patient is currently receiving or has received:

    * systemic corticosteroids within ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment. The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
    * sorivudine or brivudine within 4 weeks prior to starting capecitabine
11. Patients with concurrent severe and/or uncontrolled concurrent medical conditions that would, in the investigator's judgement, cause unacceptable safety risks, contraindicate the participation in the study or compromise compliance with the protocol (e.g., uncontrolled hypertension and/or uncontrolled diabetes mellitus, clinically significant pulmonary disease, clinically significant neurological disorder, chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.)
12. Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed
13. Participation in a prior investigational study within 30 days prior to enrolment or within 5 half-lives of the investigational product, whichever is longer
14. Patient who has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug, or who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥ 25% of the bone marrow was irradiated
15. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery)
16. Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 4.03 Grade <1 (Exception to this criterion: patients with any grade of alopecia are allowed to enter the study)
17. Patient with a Child-Pugh score B or C
18. Patient has a concurrent malignancy or malignancy within 3 years of inclusion, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer
19. Patient has a history of non-compliance to medical regimen or inability to grant consent
20. Pregnant (confirmed by a positive hCG laboratory test > 5mIU/mL) or lactating women
21. Any condition which in the investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol
22. Individuals deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose (MTD) and the recommended dose for phase 2 (RP2D) of ribociclib and capecitabine combination | From baseline to the end of cycle 1, up to 21 days
  Determination of MTD and RP2D of ribociclib and capecitabine combination, PO in a 21 day schedule (2 weeks on/1 week off), in subjects eligible to a capecitabine treatment, with locally advanced/metastatic breast cancer who failed anthracycline and taxane treatment.

SECONDARY OUTCOMES:
Evaluate safety of ribociclib and capecitabine combination | Toxicities will be assessed during the whole treatment period (6 months expected in average) followed by a 1-year post-treatment follow-up period, and reported during the visits scheduled by the study flow chart
  Toxicities are graded according to the CTCAE V4
Characterize the pharmacokinetic (PK) profile of ribociclib and capecitabine combination | From baseline to the end of cycle 1, up to 21 days
  The objective of the pharmacokinetics is to investigate the interactions between ribociclib and capecitabine
Evaluate the anti-tumor activity of ribociclib and capecitabine combination | From baseline to disease progression or death from any cause, whichever comes first, up to 18 months (estimated treatment duration average: 6 months)
  Anti-tumor activity of the ribociclib and capecitabine combination will be carried out according to RECIST criteria version 1.1.
Evaluate anti-tumor activity and safety of the ribociclib and capecitabine combination RP2D according to RH status | From baseline to disease progression or death from any cause, whichever comes first, up to 18 months (estimated treatment duration average: 6 months)
  Anti-tumor activity (At baseline and every 6 weeks) according to RECIST criteria version 1.1. and Toxicities according to the CTCAE V4
Evaluate the anti-tumor activity of ribociclib and capecitabine depending on Rb status | From baseline to disease progression or death from any cause, whichever comes first, up to 18 months (estimated treatment duration average: 6 months)
  Anti-tumor activity of the ribociclib and capecitabine combination will be carried out according to RECIST criteria version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bachelot, MD/PhD, Principal Investigator — UNICANCER
Locations (2):
- France (2):
  - Centre Leon Berard, Lyon
  - Institut de Cancérologie de l'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Unicancer official website — http://www.unicancer.fr